CLINICAL TRIAL: NCT04943094
Title: Clinical and Functional Consequences of Photodynamic Diagnosis (PDD) and Intravesical Instillation Therapy
Acronym: URODYN
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Jørgen Bjerggaard Jensen, Professor, Aarhus University Hospital
Other Study IDs: URODYN
Record Dates: First submitted 2021-06-18; First posted 2021-06-29 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Non-muscle Invasive Bladder Cancer
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- TURBT alone: Patients treated with TURBT without adjuvant instillation therapy
  Interventions: Other: Urodynamic examination
- TURBT and mitomycin C: Patients treated with TURBT followed by six adjuvant instillations with mitomycin C
  Interventions: Other: Urodynamic examination
- TURBT and bacillus Calmette-Guerin: Patients treated with TURBT followed by six adjuvant instillations with BCG
  Interventions: Other: Urodynamic examination

INTERVENTIONS:
Other: Urodynamic examination — A urodynamic examination is performed in all patients four to six weeks following TURBT and repeated six months later in order to obtain bladder function and possible changes.

SUMMARY:
The aim is to evaluate and compare treatment strategies for non-muscle invasive bladder cancer. Furthermore, the impact of intravesical instillations on bladder function will be examined by urodynamic examination both prior to and following instillation therapy.

ELIGIBILITY:
Inclusion Criteria:

* non-muscle invasive bladder tumour

Exclusion Criteria:

* more than one previous bladder tumour recurrence
* muscle invasive bladder cancer (at baseline or prior to inclusion)
* utilization of urinary catheter
* have had heart valve replacement performed
* pregnant or lactating

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with primary non-muscle invasive bladder cancer or who are diagnosed with their first or second recurrence.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in urodynamic specifics (bladder compliance, detrusor overactivity, maximal cystometric capacity) | examined at time 0 and after six months
  Obtained from the urodynamic test

CONTACTS AND LOCATIONS:
Overall Officials: Jørgen B. Jensen, DMSc, MD, Study Chair — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No